I7P-MC-DSAD Statistical Analysis Plan Version 1

A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the

Efficacy and Safety of LY3041658 in Adults with Moderate-to-Severe Hidradenitis Suppurativa

NCT04493502

Approval Date: 01-Jun-2021

# Draft Statistical Analysis Plan for Clinical Studies: I7P-MC-DSAD: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of LY3041658 in Adults with Moderate-to-Severe Hidradenitis Suppurativa

#### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries.

**Note to Regulatory Authorities:** this document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

#### LY3041658 Hidradenitis Suppuruativa

Study I7P-MC-DSAD (DSAD) is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 2 study to evaluate the efficacy and safety of LY3041658 600 mg given intravenously (IV) every 2 weeks (Q2W) in adults with moderate-to-severe HS.

Eli Lilly and Company Indianapolis, Indiana USA 46285 Protocol I7P-MC-DSAD Phase 2

Statistical Analysis Plan electronically signed and approved by Lilly on date provided below.

LY3041658 Approval Date: 01-Jun-2021 GMT

# 2. Table of Contents

| Sec | ction | Page |
|---|---|---|
| 1. | Draft Statistical Analysis Plan for Clinical Studies: I7P-MC-DSAD:<br>A Multicenter, Randomized, Double-Blind, Placebo-Controlled,<br>Phase 2 Study to Evaluate the Efficacy and Safety of LY3041658 in<br>Adults with Moderate-to-Severe Hidradenitis Suppurativa | 1 |
| 2 | Table of Contents | |
| 2. | | |
| 3. | Revision History | |
| 4. | Study Objectives | |
| 4.1 | | |
| 4.2 | | |
| 4.3 | 1 3 3 | |
| 5. | | |
| 5.1 | | |
| 5.2 | | |
| 6. | A Priori Statistical Methods | 11 |
| | 1. Statistical Hypotheses | |
| | 6.1.1. Estimands | |
| 6.2 | 1 | |
| 6.3 | | |
| | 6.3.1. Analysis Populations | |
| | 6.3.2. Definition of Baseline Measures | |
| | 6.3.3. Analysis Methods | |
| 6.4 | | |
| 6.5 | - <b>F</b> | |
| 6.6 | | |
| 6.7 | | |
| | 6.7.1. Primary Endpoint | |
| | 6.7.2. Secondary Endpoints. | |
| C | 6.7.3. Exploratory Endpoints | |
| | 1 | |
| | <ul><li>6.7.3.3. Modified Sartorius Score (mSS)</li><li>6.7.3.4. International Hidradenitis Suppurativa Severity Score</li></ul> | 10 |
| | System (IHS4) | 16 |
| | 6.7.3.5. Patient-Reported Outcomes | |
| | 6.7.3.6. Pharmacokinetic Analyses | |

| 6.7.3.7. | Immunogenicity | 17 |
|---|---|---|
| 6.8. Bioana | alytical and Pharmacokinetic/Pharmacodynamic Methods | 17 |
| 6.9. Safety | Analyses | 17 |
| 6.9.1. E | xtent of Exposure | 18 |
| 6.9.2. A | dverse Events | 18 |
| 6.9.2.1. | Serious Adverse Event Analyses | 19 |
| 6.9.2.2. | Other Significant Adverse Events | 19 |
| 6.9.3. C | linical Laboratory Evaluation | 19 |
| 6.9.4. V | ital Signs and Other Physical Findings | 20 |
| | pecial Safety Topics, including Adverse Events of Special nterest | 21 |
| 6.9.5.1. | Abnormal Hepatic Tests | |
| 6.9.5.2. | Renal Function Effects | |
| 6.9.5.3. | Infections | 22 |
| 6.9.5.4. | Allergic Reactions/Hypersensitivities | 23 |
| 6.9.5.5. | Infusion Site Reactions | 24 |
| 6.9.5.6. | Suicidal Ideation and Behavior Risk Monitoring | 24 |
| 6.10. Subgro | oup Analyses | 24 |
| 6.11. Protoc | ol Deviations | 25 |
| 6.12. Interin | n Analyses and Data Monitoring | 25 |
| 6.13. Annua | l Report Analyses | 26 |
| 6.14. Clinica | al Trial Registry Analyses | 26 |
| 7. Reference | PS | 27 |
| 8. Appendic | es | 29 |

#### **Table of Contents**

| Table | Pag | е |
|---|---|---|
| | Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure and ment, and Categorical Criteria for Weight Changes for Adults | |
| | Common Terminology Criteria for Adverse Events (CTCAE) Related to | 2. |

# **Table of Contents**

Figure Page

Figure DSAD.5.1. Schema of Study I7P-MC-DSAD, a Phase 2 study to evaluate the efficacy and safety of LY3041658 in adults with moderate-to-severe hidradenitis suppurativa. ......10

# **Table of Contents**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Lilly-Defined MedDRA Preferred Terms for Herpes Zoster | 30 |
| Appendix 2. | Lilly-Defined MedDRA Preferred Terms for Tuberculosis | 31 |
| Appendix 3. | Lilly-Defined MedDRA Preferred Terms for Potential Opportunistic 34 | Infections |

# 3. Revision History

Statistical Analysis Plan (SAP) Version 1 was approved prior to unblinding.

# 4. Study Objectives

# 4.1. Primary Objective

| Objectives | Endpoints |
|---|---|
| Primary | |
| To test the hypothesis that treatment with<br>LY3041658 is superior to placebo in inducing<br>Hidradenitis Suppurativa Clinical Response<br>(HiSCR) in adult participants with moderate-to-severe hidradenitis suppurativa (HS) | Proportion of participants achieving<br>HiSCR response at Week 16 |

# 4.2. Secondary Objectives

| Objectives | Endpoints |
|---|---|
| Secondary | |
| • To evaluate the efficacy of LY3041658 compared to placebo with respect to measures of signs and symptoms and pain in adult participants with moderate-to-severe HS | <ul> <li>Mean change from baseline to Week 16 in:</li> <li>Total number of abscesses and inflammatory nodules (AN count)</li> <li>Skin Pain – HS Numeric Rating Scale (NRS)</li> </ul> |

# 4.3. Exploratory Objectives

#### **Exploratory**

Exploratory objectives and endpoints may include the following:

- To evaluate, at various time points, the efficacy of LY3041658 compared to placebo in inducing improvements in signs and symptoms and quality of life
- To characterize the pharmacokinetics (PK) of LY3041658 and to explore relationships between LY3041658 exposure and select biomarkers and clinical efficacy endpoints
- To assess the potential development of anti-LY3041658 antibodies and their impact on the safety profile and PK of LY3041658

# 5. Study Design

# 5.1. Summary of Study Design

Study I7P-MC-DSAD (DSAD) is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 2 study to evaluate the efficacy and safety of LY3041658 600 mg given intravenously (IV) every 2 weeks (Q2W) in adults with HS.

The study duration will be up to approximately 51 weeks over 4 study periods:

Screening: a period lasting up to 35 days before Week 0 (Visit 2, baseline)

<u>Treatment Period 1</u>: a 16-week, 2-group double-blind treatment period:

• At baseline (Visit 2, Week 0), eligible participants will be randomized in a 2:1 ratio to receive either LY3041658 600 mg IV Q2W or placebo IV Q2W, starting at the baseline visit.

<u>Treatment Period 2</u>: a 20-week, single-group open-label extension period:

• Starting at Week 16, all participants, including those previously assigned to placebo, will receive LY3041658 600 mg IV Q2W until the last dosing visit.

Post-treatment follow-up: a period lasting approximately 10 weeks.

- Participants will not receive study drug in this period.
- The last dose of the study drug is given at Visit 19 (Week 34). Thus, participants will have been withdrawn from study drug for a total of 12 weeks at the last post-treatment follow-up visit (Visit 802, Week 46).

Approximately 76 patients will be screened to achieve approximately 51 participants randomized in a 2:1 ratio to one of two treatment groups:

approximately 34 participants randomized to LY3041658, and approximately 17 participants randomized to placebo.

Unscheduled visits are for participants needing rescue therapy or incision and drainage. The use of concomitant medications, including rescue therapy, is described in Section 6.5 in the protocol.

Participants who permanently discontinue the study drug early (Section 7.1 in the protocol) will undergo early termination procedures, including an early termination visit (ETV) and the post-treatment follow-up visits specified in the Schedule of Activities (SoA) (Section 1.3 in the protocol).

Figure DSAD.5.1 illustrates the study design. The blinding procedure is described in the protocol.



Figure DSAD.5.1. Schema of Study I7P-MC-DSAD, a Phase 2 study to evaluate the efficacy and safety of LY3041658 in adults with moderate-to-severe hidradenitis suppurativa.

Note: Starting at Week 16 participants who received placebo in Treatment Period 1 will receive LY3041658 600 mg IV Q2W.

Abbreviations: FD = first dose; IV = intravenous; LD = last dose; Q2W = every 2 weeks; R = randomization visit; V = visit; W = study week relative to randomization visit.

#### **5.2.** Method of Assignment to Treatment

Subjects who meet all criteria for enrollment will be randomized in a 2:1 ratio to double-blind treatment at Visit 2. Assignment to treatment groups will be determined by a computer-generated random sequence using an interactive web-response system (IWRS).

#### 6. A Priori Statistical Methods

# 6.1. Statistical Hypotheses

The study will compare LY3041658 with placebo in adults with HS. The primary study objective is to demonstrate superior efficacy of LY3041658 over placebo.

The primary comparison of interest is the proportion of participants achieving HiSCR response at Week 16.

Secondary comparisons include the mean change of AN count and Skin Pain – HS NRS from baseline to Week 16.

Efficacy comparisons will be made without regard to changes to any background therapies. No adjustments for multiplicity will be made across the efficacy assessments. Participants who discontinue the treatment or the study prior to Week 16 will be considered a nonresponder for all relevant analyses.

#### 6.1.1. Estimands

The study will compare LY3041658 with placebo in participants with HS.

The primary comparison of interest is the difference in proportion of participants who achieve HiSCR response at Week 16. The primary objective is to demonstrate superiority of LY3041658 versus placebo.

The primary comparison will be assessed using a composite estimand where the intercurrent events of premature discontinuation and use of prohibited medication are part of the response definition.



# **6.2.** Sample Size Determination

Approximately 76 patients will be screened to achieve approximately 51 participants randomized in a 2:1 ratio to one of two treatment groups:

approximately 34 participants randomized to LY3041658, and

approximately 17 participants randomized to placebo.

For all randomized patients, approximately 45 patients are expected to complete the 16 weeks treatment period to ensure the validity of the study result. This sample size provides at least 80% power to the primary endpoint of HiSCR response. This calculation is a 2-sided test for superiority of LY3041658 compared to placebo on HiSCR response rate with significance level

of 0.05 CCI

# 6.3. General Considerations

Efficacy analyses will be conducted on the Modified Intent-to-Treat (mITT) and Per-Protocol Set Population. The mITT set includes all data from all randomized participants receiving at least 1 dose of the IP according to the treatment the participants were assigned. The PPS set includes all data from all randomized participants who missed no more than 1 dose of study treatment to which they were assigned up to and including Week 14.

Safety analyses will be conducted on the Safety Population. This set includes all data from all randomized participants receiving at least 1 dose of the IP according to the treatment the participants actually received.

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, unless otherwise stated. All confidence intervals (CIs) will be given at a 2-sided 95% level. Descriptive summaries of continuous data will present the group mean, standard deviation, median, minimum, maximum, and sample size. Descriptive summaries of discrete data will report the number of participants and incidence as a frequency and as a percentage. All p-values will be rounded up to 3 decimal places.

## 6.3.1. Analysis Populations

The following populations are defined for this study:

| Population | Description |
|---|---|
| Entered | All participants who sign the informed consent form |
| Modified Intent-to-Treat (mITT) | All participants randomly assigned to study intervention and who receive at least 1 dose of study intervention. Participants will be analyzed |
| | according to the intervention to which they were assigned. |
| Per Protocol Set (PPS) | All participants randomly assigned to study intervention to which they were assigned at Week 0 and who missed no more than 1 dose of study treatment up to and including Week 14. |
| Safety | All participants randomly assigned to study intervention and who receive at least 1 dose of study intervention. Participants will be analyzed according to the intervention they actually received within each study period. |
| Pharmacokinetic (PK) Analysis | All participants randomly assigned to study intervention and who receive at least 1 dose of study intervention and have PK data available. |

#### 6.3.2. Definition of Baseline Measures

The baseline value for Treatment Period 1 is defined as the last nonmissing measurement on or before the date of first study drug administration (expected at Week 0). The baseline value for Treatment Period 2 is the last available value before Visit 10 (Week 16), the visit at which participants who previously received placebo will receive their first dose of LY3041658. Other definitions of the baseline value may be used to conduct additional supporting analyses.

#### 6.3.3. Analysis Methods

The main analysis of categorical efficacy variables and health outcomes variables will use a logistic regression analysis with treatment group in the model. The p-value and 100(1-alpha)% CI for the odds ratio from the logistic regression model are used for primary statistical inference. The difference in percentages and 100(1-alpha)% CI of the difference in percentages using the Newcombe-Wilson without continuity correction will be reported. The p-value from the Fisher's exact test will also be produced as a secondary analysis.

The main analysis for all continuous efficacy and health outcomes variables will use mixed model repeated measures (MMRM) analysis. The model will include treatment, region, baseline disease severity, visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects. An unstructured (co)variance structure will be used to model the between- and within-patient errors. If this analysis fails to converge, the heterogeneous autoregressive [ARH(1)], followed by the heterogeneous compound symmetry (CSH), followed by the heterogeneous Toeplitz (TOEPH) will be used. The Kenward-Roger method will be used to estimate the degrees of freedom. Type III tests for the least-squares means (LSM) will be used for the statistical comparison. The LSM difference, standard error, p-value and 100(1-alpha)% CI will also be reported.

Fisher's exact test will be used for the adverse events (AEs), discontinuation, and other categorical safety data for between-treatment group comparisons. Continuous vital signs, body weight, and other continuous safety variables, including laboratory variables, will be analyzed by an ANCOVA with treatment group and baseline value in the model. The significance of within-treatment group changes from baseline will be evaluated by testing whether or not the treatment group LSM changes from baseline are different from zero; the standard error for the LSM change will also be displayed. Differences in LSM will be displayed, with the p-value associated with the LSM comparison to placebo and a 95% CI on the LSM difference also provided. In addition to the LSMs for each group, the within-group p-value for the change from baseline will be displayed. Treatment-emergent high/low for categorical laboratory safety analyses will also be produced.

# 6.4. Handling of Dropouts or Missing Data

Missing data on the primary endpoint, HiSCR response, and other dichotomous endpoints will be imputed as nonresponse. As a supplementary analysis, the primary endpoint at week 16 will be imputed using the last observation prior to missingness. For other endpoints, including continuous secondary endpoints, missing data may be imputed using the last observation prior to missingness or other appropriate imputation methods.

# 6.5. Patient Disposition

A description of participant disposition will be provided, including a summary of the number and percentage of participants entered into the study, enrolled in the study, and treated, as well as the number and percentage of participants completing the study (participants who receive at least

1 dose of study drug and have at least 1 postbaseline assessment), or discontinuing (overall and by reason for discontinuation). A summary of important protocol deviations will be provided.

#### 6.6. Patient Characteristics

Demographic data are collected and reported to demonstrate that the study population represents the target patient population. A summary of baseline demographics and disease characteristics, historical diagnoses, pre-existing conditions, and prior therapies will be reported using descriptive statistics. Other participant baseline characteristics will be summarized by group as deemed appropriate.

## 6.7. Efficacy and Health Outcome Analyses

# 6.7.1. Primary Endpoint

The primary comparison of interest is the proportion of participants achieving HiSCR response at Week 16. The HiSCR (Kimball et al. 2014; Kimball et al. 2016b) is defined as at least a 50% reduction in the total abscess and inflammatory nodule count (sum of abscesses and inflammatory nodules [AN count]) with no increase in abscess count (A count) and no increase in draining fistulae count (DF count) relative to baseline.



The primary comparison to establish superiority of LY3041658 over placebo using a composite estimand where the intercurrent events of premature discontinuation and use of prohibited medication are part of the response definition. The composite endpoint will be analyzed using logistic regression on the mITT and PPS population with treatment group in the model. The treatment difference and 95% CIs will be reported.

# 6.7.2. Secondary Endpoints

Secondary comparisons of interest are the mean change from baseline to Week 16 for

- total number of abscesses and inflammatory nodules (AN count), and
- Skin Pain HS NRS.

The Skin Pain – HS Numeric Rating Scale (NRS) is a patient-administered, single-question, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "pain as bad as I can imagine." The recall period is 7 days.

An analysis of covariance (ANCOVA) model with proper link function will be used for analysis of these secondary endpoints on the mITT and PPS population. The AN count is a count data and we will use log transformation as the link function.

#### 6.7.3. Exploratory Endpoints

#### 6.7.3.1. Additional HiSCR Response Definitions

The primary endpoint will be assessed using different definitions of HiSCR response at Week 16. Specifically, the needed reduction in AN count will be modified from 50% to 75% and to 90%. The same analysis method used for the primary endpoint will be used for these exploratory analyses. The percentage of responders achieving, HiSCR50, HiSCR75, and HiSCR90, in the mITT and the PPS population will be summarized by visit and by treatment arm to which the patients were randomized at Week 0 (Visit 2). A plot of the percentage of responders over weeks will be provided.

The proportion of visits that a patient achieves HiSCR response out of the total visits the patient attends during study period 1 and 2 (Week 0 to Week 36) will be calculated as follow,

$$\frac{\text{\# of visits the patient achieves HiSCR response}}{\text{Total \# of visits the patient attends}}*100.$$

The HiSCR response is defined in Section 6.7.1 which is based on a patient's baseline values. The summary statistics of the proportion of visits achieving responses will be summarized by treatment arms to which the patients were randomized at Week 0 (Visit 2).

Moreover, the restricted mean response time (RMRT), a measure of the average time a responder stays a responder within a specified time period, will be provided up for responders at week 16 up (Visit 10) to week 36 (Visit 20) in each treatment arm, respectively. The time to loss of response in HiSCR50 is defined as >= 50% increase in AN compared to the average AN count from the 3 previous visits, and the increase was >= 3 AN from the average AN count of the 3 previous visits. Specifically, the RMRT is calculated as,

$$\sum_{k=10}^{20} \left\{ \prod_{v=10}^{k} \left( 1 - \frac{\delta_v}{R_v} \right) \right\} \times 2 \text{ weeks}$$

Where  $\delta_v$  is the number of patients who are responder at Visit 10 (week 16) but first loss response at Visit v and  $R_v$  is the number of patients who are responder at Visit 10 (week 16) and stay reponse before Visit v. The average RMRT will be summarized by treatment arm to which the patients were randomized at Week 0 (Visit 2).

#### 6.7.3.2. Lesion Counts

The mean change from baseline to Week 16 for the total number of abcesses, inflammatory nodules, draining fistulae, and abscess and inflammatory nodule (AN) will be individually summarized and assessed using ANCOVA. Moreover, we will calculate the proportion of patients that achieve 50%, 75% and 90% decreases in AN count at W12 and W16. In addition to AN reduction, the proportion of patients with disease flare will be calculated up to W16, defined as a  $\geq$ 25% increase in AN count from the baseline and  $\geq$ 2 in AN count.

#### 6.7.3.3. Modified Sartorius Score (mSS)

The mean percent change from baseline to Week 16 for the total modified Sartorius Score (mSS) will be summarized by treatment group and assessed using MMRM methods.

#### 6.7.3.4. International Hidradenitis Suppurativa Severity Score System (IHS4)

The mean percent change from baseline to Week 16 for the International Hidradenitis Suppurativa Severity Score System (IHS4) will be summarized by treatment group and assessed using MMRM methods.

#### 6.7.3.5. Patient-Reported Outcomes

Categorical variables will be analyzed using logistic regression analyses, whereas the mixed-effects model of repeated measures (MMRM) will be the method of analysis for continuous endpoints. The analyses will be based on the mITT population unless otherwise specified.

The following continuous endpoints from patient-reported outcomes will be assessed:

- Mean change from baseline to Week 16 on the Dermatology Life Quality Index (DLQI)
- Mean change from baseline to Week 16 on the Drainage Numeric Rating Scale
- Mean change from baseline to Week 16 on the Smell Numeric Rating Scale

The following categorical endpoints from patient-reported outcomes will be assessed:

- Proportion of patients responding "no symptoms" on the Patient Global Impression of Severity – 7 Days (Hidradenitis Suppurativa)
- Proportion of patients responding "much better" on the Patient Global Impression of Change – 7 Days (Hidradenitis Suppurativa)
- Proportion of patients responding "much better" or "a little better" on the Patient Global Impression of Change 7 Days (Hidradenitis Suppurativa)
- Proportion of patients with baseline skin pain NRS≥3 having a decrease in skin pain NRS≥ 30%
- Proportion of patients with baseline drainage NRS≥3 having a decrease in drainage NRS≥ 30%
- Proportion of patients with baseline smell NRS≥3 having a decrease in smell NRS≥ 30%

For patients who meet the criteria at baseline for the presence of inflammatory back pain (IBP), the following endpoints will be assessed using ANCOVA:

- Mean change from baseline to Week 16 on the weekly spinal pain numeric rating scale
- Mean change from baseline to Week 16 on the weekly nightly spinal pain numeric rating scale.

#### 6.7.3.6. Pharmacokinetic Analyses

Plasma concentrations of LY3041658 will be listed by time point using descriptive statistics and displayed graphically. Actual sampling time relative to the last dose and time deviations will be considered to determine exclusions from summary statistics and mean plots.

The data may also be analyzed using a population approach via nonlinear mixed-effects modeling (NONMEM) with the NONMEM software. The PK data from Study DSAD may be combined with data from another study in the clinical development program to improve PK parameter estimation.

#### 6.7.3.7. Immunogenicity

Frequencies and percentages will be tabulated for the following:

- participants with pre-existing ADA, and
- participants who are TE-ADA positive (TE-ADA+) to LY3041658.

Treatment-emergent ADAs are defined as those with a titer 2-fold (1 dilution) greater than the minimum required dilution if no ADAs were detected at baseline (treatment-induced ADA) or those with a 4-fold (2 dilutions) increase in titer compared with baseline if ADAs were detected at baseline (treatment-boosted ADA). For the TE-ADA+ participants, the distribution of maximum titers will be described. The frequency of neutralizing antibodies, if assessed, may also be tabulated for the TE-ADA+ participants.

The relationship between the presence of ADA and the LY3041658 concentrations and PD response to LY3041658, including safety and efficacy, may also be assessed.

## 6.8. Bioanalytical and Pharmacokinetic/Pharmacodynamic Methods

Graphical analyses to explore relationships between LY3041658 exposure and select biomarkers and clinical efficacy endpoints will be performed.

# 6.9. Safety Analyses

The general methods used to summarize safety data, including the definitions of baseline values, are described in Section 6.3.2.

Safety analyses will include data after rescue unless otherwise stated, and patients will be analyzed according to the investigational product to which they were randomized at Week 0 (Visit 2). Additional analyses may be conducted using data after rescue to systemic therapy for some safety topics such as systemic treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs). Safety analyses will take place using the safety population defined in Section 6.3.1.

Safety topics that will be addressed include the following: AEs, clinical laboratory evaluations, vital signs and physical characteristics.

Unless otherwise specified, by-visit summaries will include planned on-treatment visits. For tables that summarize events (such as AEs, categorical lab abnormalities, shift to maximum value), post-last dose follow-up data will be provided for Treatment Period 1 (Week 0 to Week 16) and Treatment Period 2 (Week 16 to Week 36) separately. For deaths and malignancies, all

available follow-up data up to the end of the study will be included. Listings will include all safety data.

For selected safety assessments, descriptive statistics may be presented for the last measure observed during post-treatment follow-up (up to 30 days after the last dose of treatment including rescue, regardless of the study period).

#### 6.9.1. Extent of Exposure

Duration of exposure (in days) to study drug will be summarized for the safety population in both Period 1 and 2 by treatment group using descriptive statistics (n, mean, SD, minimum, 1<sup>st</sup> quartile, median, 3<sup>rd</sup> quartile, maximum).

For subjects without drug interruption, the duration of exposure for each patient is the date of last dose – date of first dose +1. If subjects have drug interruption, the duration of exposure for each patient is the (Treatment end date before drug interruption – date of first dose +1) + (date of last dose – treatment re-start date +1).

#### 6.9.2. Adverse Events

Adverse events are recorded in the eCRFs. Each AE will be coded to system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA) version that is current at the time of database lock. Severity of AEs is recorded as mild, moderate, or severe.

A TEAE is defined as an event that either first occurred or worsened in severity after the first dose of study treatment and on or prior to the last visit date during the analysis period. For each event classification term, the number of participants experiencing a TEAE with that classification term will be tabulated. TEAEs will be summarized by treatment period and overall for the study.

Treatment-related TEAEs are defined as events that are indicated by the investigator on the eCRF to be related to treatment. For events that are gender-specific, the denominator and computation of the percentage will include only participants from the given gender.

Adverse events are classified based upon the MedDRA PT. The MedDRA Lowest Level Term (LLT) will be used in defining which events are treatment-emergent. The maximum severity for each LLT during the baseline period up to the first dose of the study medication will be used as the baseline. If an event with missing severity is preexisting during the baseline period, and persists during the treatment period, then the <u>baseline severity</u> will be considered mild for determining TEAE (that is, the event is treatment-emergent if the severity is coded moderate or severe postbaseline and not treatment-emergent if the severity is coded mild postbaseline). If an event occurring postbaseline has a missing severity rating, then the event is considered treatment-emergent. The day and time for events where onset is on the day of the first dose of study treatment will both be used to distinguish between pretreatment and posttreatment in order to derive treatment-emergence. Should there be insufficient data for AE start date to make this

comparison (for example, the AE start year is the same as the treatment start year, but the AE start month and day are missing), the AE will be considered treatment-emergent.

In an overview table, the number and percentage of subjects who experienced a TEAE or serious adverse event (SAE), died due to an AE, or discontinued from the study due to an AE will be summarized by treatment.

The frequency and percentages of patients with TEAEs will be summarized by treatment using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC. The frequency and percentages of patients with TEAEs by maximum severity will also be summarized by treatment using MedDRA PT nested within SOC.

Fisher's exact test will be performed to compare percentages for each LY3041658 dose group and Placebo at both the SOC and PT levels.

Listings will be presented for all AEs, all SAEs, all AEs leading to death, all AEs leading to study drug temporary interruption, and all AEs leading to discontinuation from the study.

#### 6.9.2.1. Serious Adverse Event Analyses

The number and percentage of patients who experienced an SAE (including the SAEs that led to death) during the study drug period will be summarized by treatment using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC.

#### 6.9.2.2. Other Significant Adverse Events

The number and percentage of patients who permanently discontinued from study treatment due to an AE (including AEs that led to death) during the study drug period will be summarized by treatment using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC.

Fisher's exact test will be performed to compare percentages for each LY3041658 dose group and Placebo at both the SOC and PT levels.

# 6.9.3. Clinical Laboratory Evaluation

Laboratory analyses will include planned analytes only. Planned analytes are those specified in the protocol. Summaries will be provided in both Système International (SI) and United States (US) conventional (CN) units (when different). Limits from the performing lab will be used to define low and high. Analyses of laboratory values will be produced using the measurements collected at scheduled time points. All unscheduled assessments will appear only in data listings.

• Box plots for observed values: Values at each visit (starting at randomization) will be displayed in box plots for patients who have both a baseline and a result for the specified visit. Unplanned measurements will be excluded. Original-scale data will be used for the display. These box plots will be used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries. The box plot will be a notched box for each treatment with outliers displayed, individual measurements outside

- of reference limits will also be displayed using distinct symbols overlaying the box plot, and descriptive summary statistics will be included in a table below the box plot.
- Box plots for change values: Change from baseline to each visit will be displayed in box plots for patients who have both a baseline and a result for the specified visit. Change from baseline to last observation will also be summarized and analyzed for patients who have both baseline and at least 1 postbaseline result. Baseline will be the last non-missing observation in the baseline period. The last non-missing observation in the Dosing Period will be used as the last observation. Unplanned measurements will be excluded. The box plot will be a notched box for each treatment with outliers displayed, change from baseline to last observation will be summarized within the box plot of changes (rightmost column), and descriptive summary statistics will be included in a table below the box plot, along with a p-value using the ANCOVA model containing terms for treatment and the continuous covariate of baseline measurement. Type III sums of squares will be used. The significance of within-treatment group changes from baseline will be evaluated by testing whether the treatment group LSMean changes from baseline are different from zero using a t-statistic. In addition to the LSMeans and tests, the SD, minimum, Q1, median, Q3, and maximum will be displayed.

Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin will not be included in this analysis as different ranges will be used as described in Section 6.9.5.

## 6.9.4. Vital Signs and Other Physical Findings

Vital signs and physical characteristics include systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse, weight, and BMI. Original-scale data will be analyzed. When these parameters are analyzed as continuous numerical variables, unplanned measurements will be excluded. When these parameters are analyzed as categorical outcomes and/or treatment-emergent abnormalities, planned and unplanned measurements will be included.

The planned analyses described for the laboratory analytes in Section 6.9.3 will be used to analyze the vital signs and physical characteristics, except for the inclusion of a threshold for change in addition to a limit for the definition of treatment-emergent. defines the low and high baseline values as well as the criteria used to define treatment-emergence based on post-baseline values.

Table DSAD.6.1. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure and Pulse Measurement, and Categorical Criteria for Weight Changes for Adults

| | Low | High |
|---|---|---|
| Parameter | mmHg | mmHg |
| Systolic BP (mm Hg) | | |
| (Supine or sitting – | ≤90 and decrease from baseline ≥20 | ≥140 and increase from baseline ≥20 |
| forearm at heart level) | | |
| Diastolic BP (mm Hg) | | |
| (Supine or sitting – | ≤50 and decrease from baseline ≥10 | ≥90 and increase from baseline ≥10 |
| forearm at heart level) | | |

| Pulse (bpm) (Supine or sitting) | <50 and decrease from baseline ≥15 | >100 and increase from baseline ≥15 |
|---|---|---|
| Weight (kg) (Consistent clothing and timing in relationship to meals and voiding) | (Loss) decrease ≥7% | (Gain) increase ≥7% |

# 6.9.5. Special Safety Topics, including Adverse Events of Special Interest

In addition to general safety parameters, safety information on specific topics of special interest will also be presented. Additional special safety topics may be added as warranted.

In general, for topics regarding safety in special groups and circumstances, patient profiles and/or patient listings, where applicable, will be provided when needed to allow medical review of the time course of cases/events, related parameters, patient demographics, study drug treatment and meaningful concomitant medication use. In addition to the safety topics for which provision or review of patient data is specified, these will be provided when summary data are insufficient to permit adequate understanding of the safety topic.

#### 6.9.5.1. Abnormal Hepatic Tests

Analyses for abnormal hepatic tests will involve 4 laboratory analytes: ALT, AST, total bilirubin, and ALP. In addition to the analyses described in Section 6.9.3, this section describes specific analyses for this topic.

The central laboratory reference ranges (CLRM reference ranges) will be used for these laboratory assessments (ALT, AST, total bilirubin, and ALP).

Analyses for change from baseline to last observation, change from the baseline value to the minimum value during Period 1 and 2, change from the baseline value to the maximum value during Period 1 and 2, and treatment-emergent high or low laboratory results at any time are described in Section 6.9.3

The patients with the following abnormal elevations in hepatic laboratory tests at any time will be listed for both Period 1 and 2:

- ALT measurement  $\geq 3$  times,  $\geq 5$  times and  $\geq 10$  times the central laboratory ULN.
- AST measurement  $\geq 3$  times,  $\geq 5$  times and  $\geq 10$  times the central laboratory ULN.
- Total bilirubin measurement  $\geq 2$  times the central laboratory ULN.
- ALT or AST measurement ≥3 times the central laboratory ULN and total bilirubin measurement ≥2 times the central laboratory ULN
- ALP measurement  $\geq 2$  times the central laboratory ULN.

#### 6.9.5.2. Renal Function Effects

Effects on renal function will be assessed through analysis of elevated creatinine.

The CTCAE will be applied for laboratory tests related to renal effects (Table DSAD.6.2). This CTCAE grading scheme is consistent with both Version 3.0 and Version 4.03 of the CTCAE guidelines.

Shift tables will show the number and percentage of subjects from baseline to maximum during Period 1 and 2, with baseline depicted by highest grade during the baseline period. A shift table summary displaying the number and percentage of subjects with maximum postbaseline results will be presented by treatment group within the following categories:

- Decreased; postbaseline category < baseline category
- Increased; postbaseline category > baseline category
- Same; postbaseline category = baseline category.

Treatment-emergent lab abnormalities related to elevated creatinine occurring at any time during the Dosing Period will be tabulated using the CTCAE grades shown in Table DSAD.6.2. Planned and unplanned measurements will be included.

Treatment-emergence will be characterized using 5 criteria:

- any increase in postbaseline CTCAE grade from worst baseline grade
- increase to Grade 1 or above at worst postbaseline
- increase to Grade 2 or above at worst postbaseline
- increase to Grade 3 or above at worst postbaseline
- increase to Grade 4 at worst postbaseline.

Table DSAD.6.2 Common Terminology Criteria for Adverse Events (CTCAE) Related to Renal Effects

| Lab Test | CTCAE Version | Grade | Criteria in SI or CN Units |
|---|---|---|---|
| Elevated creatinine | 3.0 | 0 (normal) | $\leq$ ULN |
| | | 1 | > ULN and ≤1.5× ULN |
| | | 2 | $>1.5 \times$ ULN and $\leq 3 \times$ ULN |
| | | 3 | >3× ULN and ≤6× ULN |
| | | 4 | >6× ULN |

Abbreviations: CN = conventional (US); CTCAE = Common Terminology Criteria for Adverse Events; SI = Système International; ULN = upper limit of normal.

#### 6.9.5.3. Infections

Infections will be defined using the PTs from the MedDRA Infections and Infestations SOC, with additional terms from the Investigations SOC being used in selected instances, as described below.

Treatment-emergent infections will be analyzed according to various groups of infectious events including:

- all infections
  - o all PTs in the Infections and Infestations SOC.
- serious infections
  - o all PTs in the Infections and Infestations SOC that are SAEs,

- infections that require therapeutic intervention (antibiotics, antivirals, antifungals, and so on)
  - o all PTs in the Infections and Infestations SOC for which there is an antimicrobial concomitant medication associated with that event for that subject,
- herpes zoster
  - o specific Lilly-defined PTs from the Herpes Viral Infections high-level term (HLT) in the Infections and Infestations SOC, shown in Appendix 1,
- tuberculosis
  - specific Lilly-defined PTs from the Tuberculous Infections HLT and the Investigations SOC, shown in Appendix 2
- viral hepatitis
  - o all PTs from the Hepatitis Viral Infections HLT (HLT code 10057212) in the Infections and Infestations SOC.

For each infection event, the frequency for each PT will be provided, ordered by decreasing frequency in the LY3041658 highest dose group by infection group: all infections, serious infections (overall and on each approach to identifying SAEs), infections that require therapeutic intervention, herpes zoster infections, tuberculosis, and viral hepatitis.

In addition to the incidence of infectious AEs by MedDRA PT as described above, the number and percentage of subjects with treatment-emergent infectious AEs by treatment group will be summarized and listed.

#### Potential Opportunistic Infections:

Potential opportunistic infections (POIs) will be identified according to 2 different approaches.

POIs are identified from TEAEs based on a Lilly-defined list of MedDRA PTs, shown in the Appendix 3. These PTs are a subset of terms from the Infections and Infestations SOC.

For the POIs identified from MedDRA PTs, the number and percentage of subjects overall and for each specific PT will be summarized by treatment group, with specific event terms ordered by decreasing frequency in the LY3041658 highest dose.

#### Association of Infections with Lymphopenia or Neutropenia:

The relationship between the occurrence of lymphopenia and neutropenia with the occurrence of infections will be evaluated based on case reviews. Inferential analyses and/or graphical displays may be conducted if warranted. Infection outcomes considered for this analysis are any infection, any serious infection, infections that require therapeutic intervention (antibiotics, antivirals, antifungals, and so on), tuberculosis, herpes zoster, and viral hepatitis.

#### 6.9.5.4. Allergic Reactions/Hypersensitivities

A search will be performed using the current MedDRA version 20.0 SMQs to search for relevant events, using the following queries:

- Anaphylactic reaction SMQ (20000021)
- Hypersensitivity SMQ (20000214)

• Angioedema SMQ (20000024)

Events that satisfy the queries will be listed, by temporal order within patient ID, and will include SOC, PT, SMQ event categorization including detail on the scope (narrow or broad), reported AE term, AE onset and end dates, severity, seriousness, outcome, etc.

#### 6.9.5.5. Infusion Site Reactions

Symptoms of a local infusion site reaction may include erythema, induration, pain, pruritus, and edema. If an infusion site event is reported, the adverse event will be recorded, and additional data will be provided to the sponsor in the eCRF. The number and percentage of patients having any ISR, and each Symptoms (erythema, induration, pain, pruritus, and edema) by maximum severity will be summarized by and treatment for Period 1 using the mITT population. Additionally, summaries of ISR and each Symptoms over by treatment will be provided for each visit.

#### 6.9.5.6. Suicidal Ideation and Behavior Risk Monitoring

Responses to the Columbia Suicide-Severity Rating Scale (C-SSRS) will be summarized by treatment and listed for each patient.

# 6.10. Subgroup Analyses

Subgroup analyses comparing LY3041658 to placebo will be performed on the mITT and PPS population at Week 16 for the following:

- Proportion of participants achieving HiSCR response
- Mean change from baseline to Week 16 in:
  - o Total number of abscesses and inflammatory nodules (AN count)
  - Skin Pain HS Numeric Rating Scale (NRS)

The following subgroups (but not necessarily limited to only these) will be categorized into disease-related characteristics and demographic characteristics will be evaluated:

- Gender: (Male; Female)
- Race: (Asian; Black/African American; White; or Other)
- Ethnicity: (Hispanic or Latino; and Not Hispanic or Latino)
- Region: (United States; and Australia)
- Age (<40,40-65,>65)
- Weight (<60 kg, >=60 and <100 kg, >=100 kg)
- BMI ( $<25 \text{ kg/m}^2$ , >=25 and  $<40 \text{ kg/m}^2$ , >=40 kg/m<sup>2</sup>)
- Baseline Hurley stage: II, III

Descriptive statistics will be provided for each treatment and stratum of a subgroup as outlined, regardless of sample size. The subgroup analyses for categorical outcomes will be performed using logistic regression. The model will include the categorical outcome as the dependent variable and treatment, subgroup, and treatment-by-subgroup interaction as explanatory variables. Missing data will be imputed using NRI (Section 6.4). The treatment-by-subgroup interaction comparing treatment groups will be tested at the 0.1 significance level. The p-value

from the logistic regression model will be reported for the interaction test. Response counts and percentages will be summarized by treatment for each subgroup category. The difference in percentages and 100(1-alpha)% confidence interval (CI) of the difference in percentages using the Newcombe-Wilson without continuity correction will be reported. The p-value from the Fisher's exact test will also be produced.

Additional subgroup analyses on efficacy may be performed as deemed appropriate and necessary.

#### 6.11. Protocol Deviations

Protocol deviations will be tracked by the clinical team, and their importance will be assessed by key team members during protocol deviation review meetings. A list of important protocol deviations (IPDs) will be identified.

Potential examples of deviations include patients who receive excluded concomitant therapy, significant non-compliance with study medication (<80% of assigned doses taken, failure to take study medication and taking incorrect study medication), patients incorrectly enrolled in the study, and patients whose data are questionable due to significant site quality or compliance issues. Refer to a separate document for the important protocol deviations.

The number and percentage of patients having IPD(s) will be summarized within category and subcategory of deviation by treatment group for Period 1 using the mITT population. Individual patient listings of IPDs will be provided.

# 6.12. Interim Analyses and Data Monitoring

Unblinding details are given in a separate unblinding plan.

Analysis for the primary database lock will be conducted when all participants have completed the Period 1 (or discontinued Period 1 treatment).

There are two interim analyses planned for this study:

- 1. An interim analysis on unblinded safety data will be triggered when approximately 12 patients have completed 8 weeks of treatment.
- 2. An interim analysis to assess unblinded efficacy and safety data will be triggered when approximately 21 patients have completed 12 weeks of treatment

Other interim analyses may be conducted as needed. All interim analyses will be used to support planning activities associated with the development program. No adjustment of type I error will be performed.

The assessment will be conducted by an internal assessment committee with a limited number of prespecified team members who do not have direct site contact or data entry/validation responsibilities. A limited number of pre-identified individuals may gain access to the limited unblinded data, as specified in the unblinding plan, prior to the interim or final database lock.

The assessment committee is authorized to evaluate unblinded interim efficacy and safety analyses. Study sites will receive information about interim results ONLY if they need to know for the safety of their patients.

Ongoing monitoring of safety data (including AEs, SAEs, and selected laboratory measurements) will continue throughout the study using blinded data. Interim safety analyses may be conducted to review unblinded safety data. The analyses will be conducted and reviewed by an internal assessment committee composed of personnel who do not have direct site contact or data entry/validation responsibilities.

Details of the planned interim data analyses and the assessment committee data review process are included in an assessment committee charter.

# 6.13. Annual Report Analyses

Annual report analyses, such as the Development Update Safety Report (DSUR), will be documented in a separate document.

# 6.14. Clinical Trial Registry Analyses

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements.

Analyses provided for the CTR requirements include a summary of AEs, provided as a dataset which will be converted to an XML file. Both SAEs and 'Other' AE are summarized: by treatment group, by MedDRA PT.

- An AE is considered 'Serious' whether or not it is a TEAE.
- An AE is considered in the 'Other' category if it is both a TEAE and is not serious. For each SAE and 'Other' AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term
  - o the number of events experienced.
- Consistent with www.ClinicalTrials.gov requirements, 'Other' AEs that occur in fewer than 5% of patients/patients in every treatment group may not be included if a 5% threshold is chosen (5% is the minimum threshold).
- AE reporting is consistent with other document disclosures for example, the CSR, manuscripts, and so forth.

Similar methods will be used to satisfy the European Clinical Trials Database (EudraCT) requirements.

#### 7. References

- A study to evaluate the efficacy, safety, and tolerability of guselkumab for the treatment of participants with moderate to severe hidradenitis suppurativa (HS) (NOVA). ClinicalTrials.gov website. https://clinicaltrials.gov/ct2/show/NCT03628924. Updated January 22, 2020. Accessed February 13, 2020.
- A study of efficacy and safety of two secukinumab dose regimens in subjects with moderate to severe hidradenitis suppurativa (HS) (SUNRISE). ClinicalTrials.gov website. https://clinicaltrials.gov/ct2/show/NCT03713632. Updated February 6, 2020. Accessed February 13, 2020.
- A study of efficacy and safety of two secukinumab dose regimens in subjects with moderate to severe hidradenitis suppurativa (HS). (SUNSHINE). ClinicalTrials.gov website. https://clinicaltrials.gov/ct2/show/NCT03713619. Updated November 19, 2019. Accessed February 13, 2020
- A study to evaluate the efficacy and safety of bimekizumab in study participants with moderate to severe hidradenitis suppurativa (BE HEARD I). ClinicalTrials.gov website. https://clinicaltrials.gov/ ct2/show/ NCT04242446. Updated January 27, 2020. Accessed February 13, 2020.
- A study to test the efficacy and safety of bimekizumab in study participants with moderate to severe hidradenitis suppurativa (BE HEARD II). ClinicalTrials.gov website. https://clinicaltrials.gov/ ct2/show/ NCT04242498. Updated January 27, 2020. Accessed February 13, 2020.
- Basra MK, Salek MS, Camilleri L, et al. Determining the minimal clinically important difference and responsiveness of the Dermatology Life Quality Index (DLQI): further data. *Dermatology*. 2015;230(1):27-33. https://doi.org/ 10.1159/000365390
- Columbia Lighthouse Project. The Columbia Protocol for Research. Columbia-Suicide Severity Rating Scale Scoring and Data Analysis Guide. Version 2.0. Available at: http://cssrs.columbia.edu/wp-content/uploads/ScoringandDataAnalysisGuide-for-Clinical-Trials-1.pdf. Accessed 30 January 2019.
- Hongbo Y, Thomas CL, Harrison MA, et al. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? *J Invest Dermatol*. 2005;125(4):659-664. https://doi.org/10.1111/j.0022-202X.2005.23621.x
- Hurley H. Axillary hyperhidrosis, apocrine bromhidrosis, hidradenitis suppurativa, and familial benign pemphigus: surgical approach. In: Roenigk RK, Roenigk HH, editors. *Dermatologic surgery: Principles and practice*. New York: Marcel Dekker; 1989:p 729-739.
- Kimball AB, Jemec GB, Yang M, et al. Assessing the validity, responsiveness and meaningfulness of the Hidradenitis Suppurativa Clinical Response (HiSCR) as the clinical endpoint for hidradenitis suppurativa treatment. *Br J Dermatol*. 2014;171(6):1434-1442. https://doi.org/ 10.1111/bjd.13270
- Kimball AB, Okun MM, Williams DA, et al. Two phase 3 trials of adalimumab for hidradenitis suppurativa. *N Engl J Med*. 2016a;375(5):422-434. https://doi.org/ 10.1056/NEJMoa1504370

- Kimball AB, Sobell JM, Zouboulis CC, et al. HiSCR (Hidradenitis Suppurativa Clinical Response): a novel clinical endpoint to evaluate therapeutic outcomes in patients with hidradenitis suppurativa from the placebo-controlled portion of a phase 2 adalimumab study. *J Eur Acad Dermatol Venereol*. 2016b;30(6):989-994. https://doi.org/ 10.1111/jdv.13216
- Kouris A, Platsidaki E, Christodoulou C, et al. Quality of life and psychosocial implications in patients with hidradenitis suppurativa. *Dermatology*. 2016;232(6):687-691. https://doi.org/10.1159/000453355.
- Sartorius K, Emtestam L, Jemec GB, Lapins J. Objective scoring of hidradenitis suppurativa reflecting the role of tobacco smoking and obesity. *Br J Dermatol.* 2009;161(4):831-839. https://doi.org/ 10.1111/j.1365-2133.2009.09198.x
- Sieper J, van der Heijde D, Landewé R, et al. New criteria for inflammatory back pain in patients with chronic back pain: a real patient exercise by experts from the Assessment of Spondyloarthritis International Society (ASAS). *Ann Rheum Dis.* 2009;68(6):784-788. https://doi.org/ 10.1136/ard.2008.101501
- Vekic DA, Cains GD. Hidradenitis suppurativa management, comorbidities and monitoring. *Aust Fam Physician*. 2017;46(8):584-588.
- Winthrop KL, Novosad SA, Baddley JW, et al. Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance. *Ann Rheum Dis.* 2015;74(12):2107-2116. https://doi.org/ 10.1136/annrheumdis-2015-207841
- Zouboulis CC. Hidradenitis suppurativa/acne inversa: the clinical challenge [abstract]. *Experimental Dermatology*. 2006;15(6):478. Abstract. https://doi.org/ 10.1111/j.0906-6705.2006.0436a.x
- Zouboulis CC, Desai N, Emtestam L, et al. European S1 guideline for the treatment of hidradenitis suppurativa/acne inversa. *J Eur Acad Dermatol Venereol*. 2015;29(4):619-644. https://doi.org/ 10.1111/jdv.12966
- Zouboulis CC, Tzellos T, Kyrgidis A, et al. Development and validation of the International Hidradenitis Suppurativa Severity Score System (IHS4), a novel dynamic scoring system to assess HS severity. *Br J Dermatol.*. 2017;177(5):1401–1409. https://doi.org/ 10.1111/bjd.15748

# 8. Appendices

# Appendix 1. Lilly-Defined MedDRA Preferred Terms for Herpes Zoster

| Preferred Term (MedDRA Version 18.0) | Preferred Term Code |
|--------------------------------------|---------------------|
| Herpes zoster | 10019974 |
| Ophthalmic herpes zoster | 10030865 |
| Herpes zoster infection neurological | 10061208 |
| Herpes zoster oticus | 10063491 |
| Herpes zoster disseminated | 10065038 |
| Genital herpes zoster | 10072210 |
| Herpes zoster pharyngitis | 10074245 |
| Herpes zoster meningoencephalitis | 10074248 |
| Herpes zoster meningomyelitis | 10074251 |
| Herpes zoster meningitis | 10074259 |
| Herpes zoster cutaneous disseminated | 10074297 |
| Varicella zoster virus infection | 10075611 |

# Appendix 2. Lilly-Defined MedDRA Preferred Terms for Tuberculosis

| Adrenal gland tuberculosis 10001358 | Preferred Term (MedDRA Version 18.0) | Preferred Term Code |
|---|---|---|
| Bovine tuberculosis | Adrenal gland tuberculosis | 10001358 |
| Choroid tuberceles 10008779 Congenital tuberculosis 10010657 Conjunctivitis tuberculous 10010754 Cutaneous tuberculosis 10011684 Disseminated tuberculosis 10014027 Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10072568 Joint tuberculosis 1005367 Latent tuberculosis 1005367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025143 Meningitis tuberculosis 10061234 Meningitis tuberculosis 10061234 Meningitis tuberculosis 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculosis 10030200 Pericarditis tuberculosis 10066927 | Bone tuberculosis | 10056377 |
| Congenital tuberculosis 10010657 Conjunctivitis tuberculous 10010754 Cutaneous tuberculosis 10011684 Disseminated tuberculosis 10013453 Ear tuberculosis 10014027 Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10075268 Joint tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10025183 Male genital tract tuberculosis complex test positive 10070325 Oesophogeal tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Peritoneal tuberculosis 10030200 Peritoneal tuberculos | Bovine tuberculosis | 10006049 |
| Conjunctivitis tuberculosis 10010754 Cutaneous tuberculosis 10011684 Disseminated tuberculosis 10013453 Ear tuberculosis 10014027 Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10055067 Latent tuberculosis 10025143 Lymph node tuberculosis 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10025183 Male genital tract tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10055069 Pulmonary tuberculosis | Choroid tubercles | 10008779 |
| Cutaneous tuberculosis 10011684 Disseminated tuberculosis 10013453 Ear tuberculosis 10014027 Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10025183 Male genital tract tuberculosis 1002134 Meningitis tuberculosis 10070325 Oesophogeal tuberculosis 1003200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 1003200 Pericarditis tuberculous 10064743 Pulmonary tuberculosis 10037440 Renal tuberculosis 10037440 | Congenital tuberculosis | 10010657 |
| Disseminated tuberculosis 10013453 Ear tuberculosis 10014027 Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10056367 Latent tuberculosis 10025143 Lymph node tuberculosis 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 1002183 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 1005443 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculosis 10038534 </td <td>Conjunctivitis tuberculous</td> <td>10010754</td> | Conjunctivitis tuberculous | 10010754 |
| Ear tuberculosis 10014027 Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 1003583 Prostatitis tuberculoma 10066927 Pulmonary tuberculoma 10038534 Salpingitis tuberculosis 10038534 Salpingitis tuberculosis 10038534 Salpingitis tuberculosis 100386876< | Cutaneous tuberculosis | 10011684 |
| Epididymitis tuberculous 10015004 Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculosis 10037440 Renal tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculosis 10038534 Salpingitis tuberculosis 1004640 | Disseminated tuberculosis | 10013453 |
| Erythema induratum 10015213 Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10053569 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculosis 10037440 Renal tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculosis 10038534 Salpingitis tuberculosis 1004640 Thyroid tuberculosis 10044728 | Ear tuberculosis | 10014027 |
| Extrapulmonary tuberculosis 10064445 Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10070325 Oesophogeal tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculosis 10038534 Salpingitis tuberculosis 1003874 Tuberculosis 10043774 Tuberculosis 10044728 Tuberculosis 10052883 | Epididymitis tuberculous | 10015004 |
| Female genital tract tuberculosis 10061150 Immune reconstitution inflammatory syndrome associated tuberculosis 10072797 Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10070325 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10038876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10052883 Tuberculosis 10044728 Tuberculosis abscess central nervous system 100 | Erythema induratum | 10015213 |
| Immune reconstitution inflammatory syndrome associated tuberculosis Interferon gamma release assay positive Intestinal tuberculosis Joint tuberculosis Latent tuberculosis Lupus vulgaris Lupus vulgaris Lymph node tuberculosis Male genital tract tuberculosis Meningitis tuberculosis Mycobacterium tuberculosis complex test positive Oesophogeal tuberculosis Pericarditis tuberculosis Prostatitis tuberculosis Prostatitis tuberculosis Pulmonary tuberculosis Salpingitis tuberculous Salpingitis tuberculosis Spleen tuberculosis 10037440 Thyroid tuberculosis Tuberculoma of central nervous system 10052884 Tuberculous abscess central nervous system 10052884 | Extrapulmonary tuberculosis | 10064445 |
| Interferon gamma release assay positive 10072866 Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculosis 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10039463 Silicotuberculosis 10048876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculoma of central nervous system 10052883 Tuberculous abscess central nervous system 10052884 | Female genital tract tuberculosis | 10061150 |
| Intestinal tuberculosis 10075268 Joint tuberculosis 10056367 Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10038534 Salpingitis tuberculosis 10048676 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculim test positive 10044728 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Immune reconstitution inflammatory syndrome associated tuberculosis | 10072797 |
| Joint tuberculosis | Interferon gamma release assay positive | 10072866 |
| Latent tuberculosis 10065048 Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10039463 Silicotuberculosis 10049463 Silicotuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculosis 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Intestinal tuberculosis | 10075268 |
| Lupus vulgaris 10025143 Lymph node tuberculosis 10025183 Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculosis 10052883 Tuberculosis 10052883 Tuberculosi abscess central nervous system 10052884 | Joint tuberculosis | 10056367 |
| Lymph node tuberculosis Male genital tract tuberculosis 10061234 Meningitis tuberculosis 10027259 Mycobacterium tuberculosis complex test positive 10070325 Oesophogeal tuberculosis 10030200 Pericarditis tuberculosis 10055069 Peritoneal tuberculosis 10063583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10039463 Silicotuberculosis 100439463 Silicotuberculosis 10043774 Tuberculosis 10044728 Tuberculoma of central nervous system 10052884 | Latent tuberculosis | 10065048 |
| Male genital tract tuberculosis10061234Meningitis tuberculosis10027259Mycobacterium tuberculosis complex test positive10070325Oesophogeal tuberculosis10030200Pericarditis tuberculous10055069Peritoneal tuberculosis10053583Prostatitis tuberculous10064743Pulmonary tuberculoma10066927Pulmonary tuberculosis10037440Renal tuberculosis10038534Salpingitis tuberculous10039463Silicotuberculosis10048876Spleen tuberculosis10041640Thyroid tuberculosis10043774Tuberculin test positive10044728Tuberculoma of central nervous system10052883Tuberculous abscess central nervous system10052884 | Lupus vulgaris | 10025143 |
| Meningitis tuberculosis10027259Mycobacterium tuberculosis complex test positive10070325Oesophogeal tuberculosis10030200Pericarditis tuberculous10055069Peritoneal tuberculosis10053583Prostatitis tuberculous10064743Pulmonary tuberculoma10066927Pulmonary tuberculosis10037440Renal tuberculosis10038534Salpingitis tuberculous10039463Silicotuberculosis10068876Spleen tuberculosis10041640Thyroid tuberculosis10043774Tuberculin test positive10044728Tuberculosis10052883Tuberculosis10044755Tuberculous abscess central nervous system10052884 | Lymph node tuberculosis | 10025183 |
| Mycobacterium tuberculosis complex test positive Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Male genital tract tuberculosis | 10061234 |
| Oesophogeal tuberculosis 10030200 Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10063583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculoma of central nervous system 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Meningitis tuberculosis | 10027259 |
| Pericarditis tuberculous 10055069 Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculous abscess central nervous system 10052884 | Mycobacterium tuberculosis complex test positive | 10070325 |
| Peritoneal tuberculosis 10053583 Prostatitis tuberculous 10064743 Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Oesophogeal tuberculosis | 10030200 |
| Prostatitis tuberculous 10064743 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculous abscess central nervous system 10052884 | Pericarditis tuberculous | 10055069 |
| Pulmonary tuberculoma 10066927 Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculous abscess central nervous system 10052884 | Peritoneal tuberculosis | 10053583 |
| Pulmonary tuberculosis 10037440 Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculous abscess central nervous system 10052884 | Prostatitis tuberculous | 10064743 |
| Renal tuberculosis 10038534 Salpingitis tuberculous 10039463 Silicotuberculosis 10068876 Spleen tuberculosis 10041640 Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculous abscess central nervous system 10052884 | Pulmonary tuberculoma | 10066927 |
| Salpingitis tuberculous10039463Silicotuberculosis10068876Spleen tuberculosis10041640Thyroid tuberculosis10043774Tuberculin test positive10044728Tuberculoma of central nervous system10052883Tuberculosis10044755Tuberculous abscess central nervous system10052884 | Pulmonary tuberculosis | 10037440 |
| Silicotuberculosis10068876Spleen tuberculosis10041640Thyroid tuberculosis10043774Tuberculin test positive10044728Tuberculoma of central nervous system10052883Tuberculosis10044755Tuberculous abscess central nervous system10052884 | Renal tuberculosis | 10038534 |
| Spleen tuberculosis10041640Thyroid tuberculosis10043774Tuberculin test positive10044728Tuberculoma of central nervous system10052883Tuberculosis10044755Tuberculous abscess central nervous system10052884 | Salpingitis tuberculous | 10039463 |
| Thyroid tuberculosis 10043774 Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Silicotuberculosis | 10068876 |
| Tuberculin test positive 10044728 Tuberculoma of central nervous system 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Spleen tuberculosis | 10041640 |
| Tuberculoma of central nervous system 10052883 Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Thyroid tuberculosis | 10043774 |
| Tuberculosis 10044755 Tuberculous abscess central nervous system 10052884 | Tuberculin test positive | 10044728 |
| Tuberculous abscess central nervous system 10052884 | Tuberculoma of central nervous system | 10052883 |
| · | Tuberculosis | 10044755 |
| Tubaraulasis bladdar 10044759 | Tuberculous abscess central nervous system | 10052884 |
| 1 ubel culosis biaddel 10044/38 | Tuberculosis bladder | 10044758 |
| Tuberculosis gastrointestinal 10061390 | Tuberculosis gastrointestinal | 10061390 |

| Preferred Term (MedDRA Version 18.0) | Preferred Term Code |
|-------------------------------------------|---------------------|
| Tuberculosis liver | 10058120 |
| Tuberculosis of central nervous system | 10061391 |
| Tuberculosis of eye | 10044819 |
| Tuberculosis of genitourinary system | 10044828 |
| Tuberculosis of intrathoracic lymph nodes | 10044846 |
| Tuberculosis of peripheral lymph nodes | 10044965 |
| Tuberculosis ureter | 10045026 |
| Tuberculous endometritis | 10071559 |
| Tuberculous laryngitis | 10045072 |
| Tuberculous pleurisy | 10045104 |
| Tuberculous tenosynovitis | 10059161 |

# Appendix 3. Lilly-Defined MedDRA Preferred Terms for Potential Opportunistic Infections

| Preferred Term (MedDRA Version 18.0) | Preferred Term Code |
|--------------------------------------------|---------------------|
| Candida pneumonia | 10053158 |
| Respiratory moniliasis | 10038705 |
| Gastrointestinal candidiasis | 10017938 |
| Oesophageal candidiasis | 10030154 |
| Coccidioides encephalitis | 10054214 |
| Coccidioidomycosis | 10009825 |
| Cutaneous coccidioidomycosis | 10068747 |
| Meningitis coccidioides | 10027207 |
| Cryptococcal cutaneous infection | 10054216 |
| Cryptococcal fungaemia | 10067112 |
| Disseminated cryptococcosis | 10013439 |
| Gastroenteritis cryptococcal | 10011485 |
| Meningitis cryptococcal | 10027209 |
| Neurocryptococcosis | 10068368 |
| Biliary tract infection cryptosporidial | 10067319 |
| Gastroenteritis cryptosporidial | 10017899 |
| Cytomegalovirus colitis | 10048983 |
| Cytomegalovirus duodenitis | 10049014 |
| Cytomegalovirus enteritis | 10049074 |
| Cytomegalovirus enterocolitis | 10049015 |
| Cytomegalovirus gastritis | 10049016 |
| Cytomegalovirus gastroenteritis | 10051349 |
| Cytomegalovirus gastrointestinal infection | 10052817 |
| Cytomegalovirus gastrointestinal ulcer | 10075619 |
| Cytomegalovirus hepatitis | 10011830 |
| Cytomegalovirus mucocutaneous ulcer | 10065036 |
| Cytomegalovirus myelomeningoradiculitis | 10065621 |
| Cytomegalovirus myocarditis | 10056261 |
| Cytomegalovirus oesophagitis | 10049018 |
| Cytomegalovirus pancreatitis | 10049566 |
| Cytomegalovirus pericarditis | 10056721 |
| Cytomegalovirus proctocolitis | 10049019 |
| Cytomegalovirus urinary tract infection | 10051350 |
| Disseminated cytomegaloviral infection | 10049075 |
| Encephalitis cytomegalovirus | 10014586 |